CLINICAL TRIAL: NCT07251075
Title: Clinical Performance of a Point-of-Care Creatinine Testing System in Individuals With Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Tingting Xu (Industry)
Responsible Party: Sponsor-Investigator, Tingting Xu, Regulatory Affair Supervisor, Eaglenos Sciences, Inc.
Organization: Eaglenos Sciences, Inc. (Industry)
Other Study IDs: BM15861
Record Dates: First submitted 2025-09-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Diseases; Kidney Injury, Acute
Keywords: Creatinine; Chronic kidney diseases; Kidney Injury, acute; POCT; Eaglenos
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biospecimen Description: Venous blood samples from non-dialysis-dependent kidney disease participants and healthy volunteers will be collected for comparative testing of creatinine levels using the Cobas biochemical analyzer. In addition, participants will perform self-testing using the investigational Creatinine Monitoring System with fresh finger capillary whole blood. No DNA or other genetic material will be extracted from any samples, and all samples will be retained only for the purpose of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: Cobas Group: Blood creatinine measurements are performed using the Cobas biochemical analyzer with venous plasma. The results will be compared with those obtained from the investigational Eaglenos Creatinine Test System using fingerstick capillary whole blood.
  Interventions: Diagnostic Test: Reference Creatinine Test System（Cobas c 111）
- Group 2: EG Group: Blood creatinine measurements are performed using the Eaglenos Creatinine Test System with fingerstick capillary whole blood. The results will be compared with those obtained from the Cobas biochemical analyzer using venous plasma.
  Interventions: Diagnostic Test: Investigational Creatinine Test System （EG）

INTERVENTIONS:
Diagnostic Test: Reference Creatinine Test System（Cobas c 111） — This group involves the use of the Cobas biochemical analyzer for measurement of venous plasma creatinine samples. The results obtained from Cobas will be compared with those obtained from the investigational Eaglenos Creatinine Test System to evaluate the accuracy and reliability of the investigational device. Study participant management and clinical care will not be influenced by the results of these study measurements.
  Groups: Group 1: Cobas Group
Diagnostic Test: Investigational Creatinine Test System （EG） — This group involves the use of the Eaglenos Creatinine Test System, a handheld device designed for self-testing of fingerstick capillary whole blood by laypersons with non-dialysis-dependent kidney disease. The results obtained from EG will be compared with those obtained from the Cobas biochemical analyzer to evaluate the accuracy and reliability of the investigational device. Study participant management and clinical care will not be influenced by the results of these study measurements.
  Groups: Group 2: EG Group

SUMMARY:
The goal of this clinical performance study is to evaluate the accuracy and usability of the Eaglenos Creatinine Test System（referred to as EG）, a point-of-care testing (POCT) system that consists of a handheld device and its associated creatinine test strips, intended for home use by laypersons with non-dialysis-dependent kidney disease.

The main questions it aims to answer are:

1. How consistent are creatinine measurements from the investigational creatinine test system compared with the clinical standard method?
2. How usable is the Creatinine Monitoring System for laypersons in a home setting?

Researchers will compare creatinine results obtained with the investigational creatinine test system (fingerstick capillary whole blood) to those from a Cobas biochemical analysis system（referred to as Cobas) (venous plasma) to determine whether the investigational device provides accurate and reliable measurements.

Participants will:

1. Provide a venous blood sample for comparative testing.
2. Perform self-testing using the Creatinine Monitoring System without prior training.
3. Complete a usability questionnaire about their experience with the investigational creatinine test system.

DETAILED DESCRIPTION:
This clinical performance study is designed to evaluate the accuracy and usability of the Creatinine Monitoring System under controlled conditions. Prior to study initiation, the investigational device, comparator device, and associated instruments will be verified to ensure calibration and proper function. All study personnel will undergo training on the protocol, informed consent procedures, and case report form (CRF) completion, and a kick-off meeting will be held to clarify roles and responsibilities.

Participants will be enrolled strictly according to the predefined inclusion and exclusion criteria. Each subject will be assigned blinded identification numbers, including subject numbers, tester numbers, and venous blood sample numbers, to minimize bias. Venous blood will be collected for hematocrit testing and comparator analysis. Following blood collection, layperson participants will receive the complete investigational device package, including the instructions for use (IFU) and relevant labeling, and will perform self-testing without any prior training or assistance. Self-testing will take place in a separate room to avoid influence from previous participants. Disinfection of the handheld electrochemical meter will be performed using CLOROX HEALTHCARE Bleach Germicidal Wipes as specified in the user manual.

After completing self-testing, layperson participants will assess the usability of the device by filling out a structured questionnaire, focusing on IFU readability and ease of use. In parallel, trained observers will complete an observer questionnaire to document any operational errors or deviations during the testing process.

Once all testing is complete, results will be unblinded. Study data will be collected and verified by the clinical research associate (CRA) for completeness and accuracy of the CRFs. Statistical analyses will then be performed by qualified statisticians on the finalized dataset, and findings will be summarized in a clinical performance study report.

Importantly, this study is observational in nature. The investigational and reference creatinine measurements are performed for research purposes only. Clinical diagnosis, treatment, and patient management are not affected by the investigational device results, and all medical care is provided according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal creatinine levels or suspected kidney disease;
* Aged 18 and above, gender is not limited;
* Voluntarily participate in this clinical study by signing the informed consent form.

Exclusion Criteria:

* The HCT range is not within 25-65%;
* Severe mental illness or other conditions that make the patient unable to cooperate;
* Inability to read or write in English language;
* Incomplete subject information (including but not limited to gender, age, education level, clinical diagnosis information; etc.);
* Previous experience with this creatinine monitoring system or similar self-monitoring devices (including but not limited to those for glucose, ketones, total cholesterol, etc.);
* Other conditions that, in the opinion of the investigator, make participation in this clinical trial inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Include at least 80% patients with varying stages of non-dialysis dependent kidney disease, as well as a small group (e.g.<20 %) of healthy volunteers and dialysis-dependent kidney disease patients, to cover the reference interval of the creatinine concentration. All subjects should be naive to this creatinine monitoring system and the similar self-monitoring devices (including but not limited to glucose, ketone, total cholesterol, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Creatinine Concentrations Measured by the Eaglenos Creatinine Test System Compared With the Cobas c 111 | Day 0 (at the time of blood sample collection).
  Creatinine concentrations (mg/dL) will be measured in fingerstick capillary whole blood using the Eaglenos Creatinine Test System and in venous plasma using the Cobas c 111 analyzer. Agreement between the two systems will be assessed using Bland-Altman analysis.
Correlation of Creatinine Concentrations Between the Eaglenos Creatinine Test System and the Cobas c 111 | Day 0 (at the time of blood sample collection).
  Creatinine concentrations (mg/dL) measured by the Eaglenos Creatinine Test System (capillary whole blood) and the Cobas c 111 analyzer (venous plasma) will be assessed for linear correlation using Pearson's correlation coefficient (r).
Predicted Differences in Creatinine Concentrations at Predefined Medical Decision Levels Between the Eaglenos Creatinine Test System and the Cobas c 111 | Day 0 (at the time of blood sample collection).
  Creatinine concentrations (mg/dL) measured by the Eaglenos Creatinine Test System (capillary whole blood) and the Cobas c 111 analyzer (venous plasma) will be used to calculate predicted differences (predicted bias) at predefined medical decision levels using Passing-Bablok regression based on all paired measurements. These levels correspond to clinically relevant cut-off values for patient management.
Number of Outlier Measurements in Creatinine Concentration Between the Eaglenos Creatinine Test System and Cobas c 111 | Day 0 (at the time of blood sample collection).
  Outliers in paired creatinine measurements (mg/dL) from the Eaglenos Creatinine Test System (capillary whole blood) and the Cobas c 111 analyzer (venous plasma) will be identified using the Extreme Studentized Deviate (ESD) method. The frequency of outlier values will be reported.
System Usability Score of the Eaglenos Creatinine Test System by Laypersons | Day 0 (at the time of blood sample collection).
  The overall usability of the Eaglenos Creatinine Test System will be evaluated using the System Usability Scale (SUS), a standardized questionnaire. SUS scores range from 10 (lowest usability) to 50 (highest usability), with higher scores indicating better usability. The distribution of participants across score segments will be reported.

IPD SHARING:
Plan to Share IPD: Yes
All collected lPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Data will be made available to qualified researchers upon submission of a research proposal and executionof a data use agreement. Data access will be granted after the final study results are published and after anethical review by the institution's ethics board. Data sharing will be coordinated via email. Qualifiedresearchers can contact xu_tingting@eaglenos.com to request access to the data.